CLINICAL TRIAL: NCT06497751
Title: Pilot Randomized Controlled Trial of Couple-based Intervention on Relationship Satisfaction and Quality of Life in HIV Male Serodiscordant Couples
Brief Title: Couple-based Intervention on Quality of Life in HIV Male Serodiscordant Couples
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Nancy Xiaonan Yu, Associate Professor, City University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: United together
Record Dates: First submitted 2024-07-03; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Quality of Life; Hiv; Relationship, Social
Keywords: Dyadic Coping; Serodiscordant Couples; Randomized Controlled Trial; China
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Couple-based Dyadic Coping Group (Experimental): The investigators will deliver three sessions (we-disease appraisal, communication skills, and dyadic coping skills) once per week. The first two sessions last 30 mins, and the final session lasts one hour.
  Interventions: Behavioral: Couple-based Dyadic Coping Group
- Usual Care Group (No Intervention): Participants received routine care from health providers.

INTERVENTIONS:
Behavioral: Couple-based Dyadic Coping Group — Session one: We-disease appraisal (30 minutes). Couples will work toward a congruent perception of HIV as a shared disease, enhancing illness control.
  Session two: Couple communication (30 minutes). Couples will learn basic knowledge of effective communication and undertake skill-building exercises focusing on effective communication techniques.
  Session three: Dyadic coping (60 minutes). Couples will learn basic knowledge of dyadic coping and work on skill-building exercises (e.g., three-phase dyadic coping exercise) to enhance support mobilization.
  Arms: Couple-based Dyadic Coping Group

SUMMARY:
This study aims to provide preliminary evidence of the efficacy of couple-based intervention over usual care in HIV serodiscordant couples in China. The investigators hypothesize that couple-based intervention would be more effective than usual care concerning both partners' quality of life and relationship satisfaction. The investigators also pilot the feasibility, acceptability, and appropriateness of the intervention content and implementation.

HIV serodiscordant couples in the intervention arm will receive three sessions of dyadic intervention. In contrast, couples in the control arm will receive usual care.

ELIGIBILITY:
The inclusion criteria for couples will be: (a) both partners are males, (b) both partners age over 18, (c) both partners report being a couple for at least three months, (d) one partner is HIV positive and the other partner is HIV-negative (i.e., serodiscordant couples), and (e) both partners are willing to participate.

The exclusion criteria for couples will be: (a) either partner cannot complete the assessment due to a low education level or physical or psychological constraint, and (b) either partner has been diagnosed with another life-threatening disease (e.g., cancer).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Change of Health-related Quality of Life | Baseline, one month (immediately after the last session of intervention), and two month
  Health-related quality of life will be measured using the 24-item World Health Organization Quality of Life, which contains four domains (i.e., physical, psychological, social relationships, and environment) (WHO, 1998). Both partners will answer this scale. Items are scored on a five-point scale (0-4). The total score for this scale is calculated by summing the scores for the four domains. The score range is 0-96. Higher scores indicate a higher level of quality of life.
Change of Relationship Satisfaction | Baseline, one month (immediately after the last session of intervention), and two month
  Relationship satisfaction will be assessed using the 4-item Couple Satisfaction Index (Funk &Rogger, 2007). Both partners will answer this scale. Items are scored on a six-point scale (0-5). The total score for this scale is calculated by summing all items. The score range is 0-20. Higher scores indicate a higher level of relationship satisfaction.
Perceived Acceptability, Appropriateness, and Feasibility | One month (immediately after the last session of intervention)
  Perceived acceptability, appropriateness, and feasibility will be assessed using the 12-item Implementation Outcome Inventory (Weiner et al., 2017). Only couples in the intervention group will answer this scale. Items are scored on a five-point scale (0-4). The total score for this scale is calculated by summing all items. The score range is 0-48. Higher scores indicate a higher level of acceptability, appropriateness, and feasibility.

SECONDARY OUTCOMES:
Change of We-disease Appraisal | Baseline, one month (immediately after the last session of intervention), and two month
  We-disease appraisal will measure the couples' appraisals of HIV ownership using a modified item of the Inclusion of Other in the Self Scale (Aron et al., 1992). Both partners will answer this scale. The total score is based on this single item. The score range is 0-6. Higher scores indicate a higher level of we-disease appraisal.
Change of Dyadic Coping | Baseline, one month (immediately after the last session of intervention), and two month
  Dyadic coping will be assessed using the 35-item Dyadic Coping Inventory (Bodenmann, 2008). Both partners will answer this scale. Items are scored on a five-point scale (0-4). The total score for this scale is calculated by summing all items. The score range is 0-140. Higher scores indicate a higher level of dyadic coping.
Change of Active Listening | Baseline, one month (immediately after the last session of intervention), and two month
  Active listening will be assessed using the 11-item Active-Empathetic Listening Scale (Bodie, 2011). Both partners will answer this scale. Items are scored on a seven-point scale (0-6). The total score for this scale is calculated by summing all items. The score range is 0-66. Higher scores indicate a higher level of active empathetic listening.
Change of Depressive Symptoms | Baseline, one month (immediately after the last session of intervention), and two month
  Depressive symptoms will be assessed using the 10-item Center for Epidemiologic Studies Depression Scale (Radloff, 1977). Both partners will answer this scale. Items are scored on a four-point scale (0-3). The total score for this scale is calculated by summing all items. The score range is 0-30. Higher scores indicate a higher level of depressive symptoms.
Change of Antiretroviral therapy Adherence | Baseline, one month (immediately after the last session of intervention), and two month
  Antiretroviral therapy adherence will be assessed using the 3-item Antiretroviral therapy Adherence Scale (Wilson et al., 2016). Only HIV-positive partners will answer this scale. Items are scored on a six-point scale (0-5). The total score for this scale is calculated by summing all items. The score range is 0-15. Higher scores indicate a higher level of adherence.
Change of Condom Use with Study Partner | Baseline, one month (immediately after the last session of intervention), and two month
  Condom use with study partner will be assessed using the 2-item condom use scale tailored for serodiscordant couples (Wyatt., 2010). Both partners will answer this scale. Both partners will answer the use of condoms during sex and sexual behaviors they had engaged in with study partners. The score ranges for both items are 0-30. The ratio was calculated by the number of condom use and the number of sexual behaviors in the past 30 days. Higher ratio indicate higher level of protected sex.
Change of Self-regulation in Relationship | Baseline, one month (immediately after the last session of intervention), and two month
  Self-regulation in relationship will be assessed using the 16-item Behavioral Self-regulation for Effective Relationships Scale (Wilson et al., 2005). Both partners will answer this scale. Items are scored on a five-point scale (0-4). The total score for this scale is calculated by summing all items. The score range is 0-64. Higher scores indicate a higher level of self-regulation.
Change of Well-being | Baseline, one month (immediately after the last session of intervention), and two month
  Well-being will be assessed using the 5-item WHO Well-being Index (WHO, 2004). Both partners will answer this scale. Items are scored on a six-point scale (0-5). The total score for this scale is calculated by summing all items. The score range is 0-25. Higher scores indicate a higher level of well-being.
Percentage of Couples Agreeing to Participate | Baseline
  The investigators will calculate the percentage of couples agreeing to participate.
Percentage of Couples Randomized to the Intervention Arm Completed All Three Sessions | One month (immediately after the last session of intervention)
  The investigators will calculate the percentage of couples randomized to the intervention arm completed all three sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Xiaonan Yu, PhD, Principal Investigator — City University of Hong Kong
Locations (4):
- China (4):
  - Jin Tang Six-color Rainbow Healthcare Service Center, Chengdu
  - Guangzhou Yue Le Health Service Center, Guangzhou
  - Community Always There, Shenzhen
  - Fangzhouai Garden, Xiamen

IPD SHARING:
Plan to Share IPD: No